CLINICAL TRIAL: NCT06353347
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study Evaluating the Efficacy and Safety of HTD1801 in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin
Brief Title: Efficacy and Safety of Berberine Ursodeoxycholate (HTD1801) in Patients With Type 2 Diabetes Inadequately Controlled With Metformin
Acronym: SYMPHONY-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Collaborators: Shenzhen HighTide Biopharmaceutical Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTD1801.PCT106
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTD1801 (Experimental): Administered orally twice daily (BID)
  Interventions: Drug: HTD1801
- Placebo (Placebo Comparator): Administered orally BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTD1801 — HTD1801 1000 mg administered orally BID as four capsules
  Other Names: berberine ursodeoxycholate
  Arms: HTD1801
Drug: Placebo — Matching placebo administered orally BID as four capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to evaluate the efficacy and safety of berberine ursodeoxycholate (HTD1801) compared to placebo in patients with type 2 diabetes inadequately controlled with metformin.

DETAILED DESCRIPTION:
This Phase 3, randomized, double-blind, placebo-controlled study will evaluate the safety and efficacy of HTD1801 in two phases, a 24-week double-blind phase followed by a 28-week open-label extension. To ensure stabilization of glycemic control, eligible patients will first participate in a 4-week single-blind run-in period where investigators will provide guidance on lifestyle modifications, concomitant medications, and procedures for self-monitoring of blood glucose. Following this period, patient eligibility will be reassessed. Eligible patients will then be randomized 2:1 to receive HTD1801 1000 mg twice daily (BID) or placebo for 24 weeks.

Patients who complete the double-blind treatment phase will enter an open-label extension period where all patients will receive HTD1801 1000 mg BID for 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes
* Received a stable dose of metformin monotherapy for at least 8 weeks prior to screening
* If used any glucose-lowering drugs other than metformin within the 8 weeks prior to screening such use was ≤7 days and was discontinued at least 4 weeks prior to screening
* Have HbA1c ≥7.5% to ≤11.0% (screening) and HbA1c ≥7.0% to ≤10.5% (pre-randomization)
* Have fasting plasma glucose ≤13.9 mmol/L (screening and pre-randomization)
* Have a body mass index ≥19.0 kg/m^2 to ≤35.0 kg/m^2

Exclusion Criteria:

* Have type 1 diabetes
* Have had any acute diabetic complications within 12 months prior to screening
* Have had any Grade 3 hypoglycemic event within 12 months prior to screening
* Have had proliferative retinopathy or macular degeneration, severe diabetic neuropathy, or diabetic foot
* Have been taking any weight loss medication or dietary supplement, have participated in a weight loss program, or have adhered to a special diet within 12 weeks prior to screening
* Have used insulin or an insulin analogue for more than 14 days within 12 months prior to screening
* Have used any hypoglycemic drug other than metformin during the 4-week run-in period prior to randomization
* Have had weight gain or loss ≥5% during the 4-week run-in period prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: mean change in HbA1c | 24 Weeks
  Mean change in HbA1c from baseline to Week 24

SECONDARY OUTCOMES:
Double-blind (DB) Phase: mean change in fasting plasma glucose | 24 Weeks
  Mean change in fasting plasma glucose from baseline to Week 24
DB Phase: mean change in 2-hour postprandial glucose | 24 Weeks
  Mean change in 2-hour postprandial glucose from baseline to Week 24
DB Phase: proportion of patients achieving HbA1c <7.0% | 24 Weeks
  Proportion of patients achieving HbA1c target value of <7.0% at Week 24
DB Phase: proportion of patients achieving HbA1c <6.5% | 24 Weeks
  Proportion of patients achieving HbA1c target value of <6.5% at Week 24
DB Phase: mean change in insulin sensitivity (HOMA-IR) | 24 Weeks
  Mean change in homeostatic model Assessment for insulin resistance (HOMA-IR) from baseline to Week 24
DB Phase: mean change in low-density lipoprotein cholesterol (LDL-C) | 24 Weeks
  Mean change in LDL-C from baseline to Week 24

OTHER OUTCOMES:
Open-Label Extension (OLE) Phase: mean change in HbA1c | 52 Weeks
  Mean change HbA1c from baseline to Week 52
OLE Phase: mean change in 2-Hour postprandial glucose | 52 Weeks
  Mean change in 2-Hour postprandial glucose from baseline to Week 52
OLE Phase: proportion of patients achieving HbA1c <7.0% | 52 Weeks
  Proportion of patients achieving HbA1c target value of <7.0% at Week 52
OLE Phase: proportion of patients achieving HbA1c <6.5% | 52 Weeks
  Proportion of patients achieving HbA1c target value of <6.5% at Week 52
OLE Phase: mean change in insulin sensitivity (HOMA-IR) | 52 Weeks
  Mean change in HOMA-IR from baseline to Week 52
OLE Phase: mean change in LDL-C | 52 Weeks
  Mean change in LDL-C from baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Kui Liu, MD, Study Director — Shenzhen HighTide Biopharmaceutical Ltd.
Locations (64):
- China (64):
  - Baogang Hospital of Inner Mongolia, Baotou
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Luhe Hospital Capital Medical University, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The Second Norman Bethune Hospital of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - Hunan Provincial People's Hospital, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Chongqing University Three Gorges Hospital, Chongqing
  - The Third People's Hospital of Datong, Datong
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Handan First Hospital, Handan
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Hospital, Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - Hengshui People's Hospital (Harrison International Peace Hospital), Hengshui
  - Heze Municipal Hospital, Heze
  - Huai'an First People's Hospital, Huai'an
  - Huangshi Central Hospital, Huangshi
  - Huizhou Municipal Central Hospital, Huizhou
  - Huzhou Central Hospital, Huzhou
  - Jinan Central Hospital, Jinan
  - Jingzhou Central Hospital, Jingzhou
  - Jinzhou Central Hospital, Jinzhou
  - The First People's Hospital of Kashgar, Kashgar
  - Hebei Petro China Center Hospital, Langfang
  - Liaocheng People's Hospital, Liaocheng
  - The First Affiliated Hospital of Henan University of Science and Technology (Jinghua), Luoyang
  - The First Affiliated Hospital of Henan University of Science and Technology (Kaiyuan), Luoyang
  - Nanjing Drum Tower Hospital - The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Nanjing First Hospital, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - Sir Run Run Hospital Nanjing Medical University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The First People's Hospital of Nanning, Nanning
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Panjin Liaohe Oilfield Gem Flower Hospital, Panjin
  - The First Hospital of Qiqihar, Qiqihar
  - Shanghai East Hospital of Tongji University, Shanghai
  - Shanghai Pudong New Area People's Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The Sixth People's Hospital of Shenyang, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen
  - Taihe Hospital, Shiyan
  - Siping City Central People's Hospital, Siping
  - The First Affiliated Hospital of Suzhou University, Suzhou
  - People's Hospital of Tianjin, Tianjin
  - Tonghua Central Hospital, Tonghua
  - The Central Hospital of Wuhan, Wuhan
  - Yijishan Hospital of Wannan Medical College, Wuhu
  - The First People's Hospital of Xiangtan City, Xiangtan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Yanan University Affiliated Hospital, Yanan
  - Yueyang People's Hospital, Yueyang
  - Yuncheng Central Hospital, Yuncheng
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
  - Zhumadian Central Hospital, Zhumadian
  - Zhuzhou Central Hospital, Zhuzhou
  - Zibo Central Hospital, Zibo
  - The First People's Hospital of Zunyi, Zunyi

IPD SHARING:
Plan to Share IPD: No